CLINICAL TRIAL: NCT06261658
Title: Improving the Quality of Cryopreserved Ovarian Tissue Reimplantation Using Platelet-enriched Autologous Plasma
Acronym: TESOVA2022
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Renato Seracchioli, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESOVA2022
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cryopreservation; Ovary Injury; Infertility, Female; Menopause Ovarian Failure
Keywords: Cryopreserved Ovarian Tissue; Ovarian tissue transplantation; Platelet-enriched Autologous Plasma; ovarian endocrine function; livebirths
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Cryopreserved Ovarian Tissue Reimplantation Using Platelet-enriched Autologous Plasma
  Interventions: Procedure: Cryopreserved Ovarian Tissue Reimplantation

INTERVENTIONS:
Procedure: Cryopreserved Ovarian Tissue Reimplantation — Cryopreserved Ovarian Tissue Reimplantation Using Platelet-enriched Autologous Plasma

SUMMARY:
The study is aimed to evaluate the effects of intraovarian injection of autologous Platelet-enriched Autologous Plasma on the outcomes of orthotopic transplantation of cryopreserved ovarian tissue.

ELIGIBILITY:
Inclusion Criteria:

* request for cryopreserved ovarian tissue transplantation;
* premature ovarian failure or irregular mentrual cycles;
* negative test for HIV, HBV, HCV, Treponema pallidum;
* negative PAP test;
* oncological authorization;
* absence of neoplastic contamination in the cryopreserved ovarian tissue;
* Informed consent

Exclusion Criteria:

* neoplastic contamination in cryopreserved ovarian tissue;
* history of endometriosis;
* endocrinological disorders present and not treated (uncompensated thyroid dysfunction, diabetes (type 1, type 2);
* body mass index (BMI) >30 kg/m2;
* circulating platelet level < 150,000 / mml;
* bacterial infection;
* ongoing use of anticoagulants;
* bleeding diathesis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-29 (Estimated); Study Completion 2033-12-29 (Estimated)

PRIMARY OUTCOMES:
Safety of Cryopreserved ovarian tissue transplantation Using Platelet-enriched Autologous Plasma | first year
  to evaluate the safety of intraovarian PRP injection in terms of absence of adverse reactions to laparoscopic ovarian tissue reimplantation surgery. Patients in early menopause or with irregular menstrual cycles who have cryopreserved their ovarian tissue at the Cryobank of Division of Gynaecology and Human Reproduction Physiopathology, IRCCS Azienda Ospedaliero-Universitaria di Bologna will be recruited. These patients will be joined by a historical cohort of patients who have the inclusion criteria of this study and who have already undergone reimplantation of ovarian tissue as the routine clinical care procedure.

SECONDARY OUTCOMES:
Effectiveness of Cryopreserved ovarian tissue transplantation Using Platelet-enriched Autologous Plasma | 9 years
  to evaluate whether the use of autologous PRP during the ovarian tissue transplantation leads to an improvement of outcomes in terms of ovarian function recovery (endocrine and reproductive functions). Patients in early menopause or with irregular menstrual cycles who have cryopreserved their ovarian tissue at the Cryobank of Division of Gynaecology and Human Reproduction Physiopathology, IRCCS Azienda Ospedaliero-Universitaria di Bologna will be recruited. These patients will be joined by a historical cohort of patients who have the inclusion criteria of this study and who have already undergone reimplantation of ovarian tissue as the routine clinical care procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Study Chair — IRCCS AOU Bologna
Locations (1):
- Diego Raimondo, Bologna, BO, Italy

REFERENCES:
- [Background] Petryk N, Petryk M. Ovarian Rejuvenation Through Platelet-Rich Autologous Plasma (PRP)-a Chance to Have a Baby Without Donor Eggs, Improving the Life Quality of Women Suffering from Early Menopause Without Synthetic Hormonal Treatment. Reprod Sci. 2020 Nov;27(11):1975-1982. doi: 10.1007/s43032-020-00266-8. Epub 2020 Jul 22. PMID 32700285
- [Background] Bos-Mikich A, de Oliveira R, Frantz N. Platelet-rich plasma therapy and reproductive medicine. J Assist Reprod Genet. 2018 May;35(5):753-756. doi: 10.1007/s10815-018-1159-8. Epub 2018 Mar 21. PMID 29564738
- [Background] Mouanness M, Ali-Bynom S, Jackman J, Seckin S, Merhi Z. Use of Intra-uterine Injection of Platelet-rich Plasma (PRP) for Endometrial Receptivity and Thickness: a Literature Review of the Mechanisms of Action. Reprod Sci. 2021 Jun;28(6):1659-1670. doi: 10.1007/s43032-021-00579-2. Epub 2021 Apr 22. PMID 33886116
- [Background] Sharara FI, Lelea LL, Rahman S, Klebanoff JS, Moawad GN. A narrative review of platelet-rich plasma (PRP) in reproductive medicine. J Assist Reprod Genet. 2021 May;38(5):1003-1012. doi: 10.1007/s10815-021-02146-9. Epub 2021 Mar 15. PMID 33723748
- [Background] Seckin S, Ramadan H, Mouanness M, Kohansieh M, Merhi Z. Ovarian response to intraovarian platelet-rich plasma (PRP) administration: hypotheses and potential mechanisms of action. J Assist Reprod Genet. 2022 Jan;39(1):37-61. doi: 10.1007/s10815-021-02385-w. Epub 2022 Feb 17. PMID 35175511
- [Derived] Ferla S, Fucina S, Clemente N, Spessotto P, Cannizzaro R, Ditto A. Probe-Based Confocal Laser Endomicroscopy in Gynecologic Surgical Oncology: Intraoperative Insights to Guide Surgical Resection. Ann Surg Oncol. 2026 Jan 14. doi: 10.1245/s10434-025-19055-1. Online ahead of print. PMID 41535563